CLINICAL TRIAL: NCT00029406
Title: Transfusion Infections Pediatric Prospective Study (TRIPPS)
Acronym: TRIPPS
Status: Completed | Type: Observational
Sponsor: Naomi Luban (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor-Investigator, Naomi Luban, MD, Children's National Research Institute
Organization: Children's National Research Institute (Other)
Other Study IDs: 990; R01HL067229 (NIH)
Record Dates: First submitted 2002-01-10; First posted 2002-01-11 (Estimated); Last update posted 2015-12-16 (Estimated); Status verified 2015-12

CONDITIONS: Blood Donors; Blood Transfusion; Cytomegalovirus Infections; Hepatitis, Viral, Human; HIV Infections
MeSH Terms: conditions — Cytomegalovirus Infections; Hepatitis, Viral, Human; HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood and plasma samples
Oversight: Data Monitoring Committee: No

SUMMARY:
To conduct a prospective study of pediatric transfusion recipients to determine the risk of transmitting various infectious agents by blood transfusion.

DETAILED DESCRIPTION:
BACKGROUND:

Despite a marked reduction in the risk of transfusion-transmitted disease, lessons learned from the delayed recognition of HIV transmission by transfusion, underscore the necessity for continued vigilance for blood safety. The study will correct a significant lack of prospective studies of transfusion transmitted disease in infants and children in this country. A critical material outcome of the study will be the establishment of a large serum and cell repository of linked patient recipient samples. Such a repository, representing prospective studies in a pediatric population, will be unique. It will provide a means for ongoing surveillance to identify more rapidly emerging infectious agents and to aid in determining whether they present a significant risk to the blood supply. Because of a close collaboration and parallel structure with two related adult transfusion studies, age related comparisons of viral clearance and clinical outcomes should likewise be derived from this work.

DESIGN NARRATIVE:

The prospective study of pediatric transfusion recipients will determine the residual risk of transmitting known infectious agents such as hepatitis viruses, human immunodeficiency virus (HIV) and human T-cell leukemia virus (HTLV), for which there are current donor screening assays, and the potential risk of known agents that are not routinely screened during blood donation, but might, nonetheless, infect blood recipients with diseases such as cytomegalovirus, parvovirus B-19, human herpes virus-8 (HHV-8) and newly proposed hepatitis viruses, TTV and the SEN virus (SEN-V). An additional primary goal of the study is to establish a repository of linked donor and recipient samples so that if a new infectious agent emerges in the future, testing of the repository will rapidly establish whether or not that agent presents a threat to the blood supply.

To insure larger numbers of samples and greater statistical power, samples from this study will be merged into a large repository to be generated in the NHLBI-sponsored RADAR (REDS Allogeneic Donor and Recipient) study. The current study will be the only pediatric arm of the RADAR multi-center study. Further, the current pediatric study will be undertaken collaboratively with a similarly designed study in adults being conducted at the NIH Clinical Center. In both studies recipients will be enrolled prior to transfusion and then followed for at least 6 months post-transfusion. Blood samples will be obtained before and at 2, 4, 8, 12, 16 and 24 weeks after transfusion. Molecular and serologic testing will be routinely performed for the agents cited above with particular emphasis on molecular assays for human retroviruses (HRV), hepatitis C virus (HCV). HIV, SEN-V, cytomegalovirus (CMV), parvovirus B-i 9 and human herpesvirus-8 (HHV-8). Aliquots will be retained in frozen storage. In addition, pre and post-transfusion and donor whole blood samples will be frozen to allow for recovery of recipient DNA and identification of microchimerism. Such microchimerism may result in transfusion-associated graft versus host disease and immunosuppression and have long term consequences for the development of immune mediated diseases in the recipient. In summary, the primary pediatric study and the proposed collaborations will allow for determinations of the transfusion risk of a variety of blood-screened and unscreened infectious agents, and will allow for comparisons of transfusion risk between pediatric and adult patients, as well as comparisons of viral persistence and clinical outcome according to age. In addition, by contributing pre and post-transfusion samples from blood recipients and their linked donor samples, this study will help establish a large serum and cell repository that will allow for the future determination of whether virtually any infectious agent is transfusion-transmitted and a potential risk to blood recipients.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric cardiac, orthopedic, and neurosurgery patients
* Trauma patients who are transfused
* Sickle cell patients who are sporadically transfused
* No allogeneic transfusion in the 6 weeks preceding the index transfusion
* A pre-transfusion sample is available from the recipient
* Life expectancy greater than 6 months
* Residence in the continental US

Exclusion Criteria:

* History of allogeneic blood transfusion in the prior three months
* Currently pregnant
* Patients on dialysis
* Patients with conditions causing significant immunosuppression

Ages: 6 Months to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Pediatric recipients of allogeneic blood transfusion and linked blood donors
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2001-04; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Rates of transfusion-transmitted viruses | 6 months post-transfusion

SECONDARY OUTCOMES:
Prevalence of newly emerging transfusion-transmitted viruses in blood donors | 6 months post-transfusion

CONTACTS AND LOCATIONS:
Overall Officials: Naomi Luban, Principal Investigator — Children's National Research Institute

REFERENCES:
- [Background] Wong EC, Perez-Albuerne E, Moscow JA, Luban NL. Transfusion management strategies: a survey of practicing pediatric hematology/oncology specialists. Pediatr Blood Cancer. 2005 Feb;44(2):119-27. doi: 10.1002/pbc.20159. PMID 15452914